CLINICAL TRIAL: NCT03467997
Title: Effects of Mental Stress and Diesel Exhaust on Cardiovascular Health
Brief Title: Mental Stress & Diesel Exhaust on Cardiovascular Health
Acronym: DESTRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Anjum Hajat, Assistant Professor, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: STUDY00002051; R00ES023498 (NIH)
Record Dates: First submitted 2017-12-12; First posted 2018-03-16 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Blood Pressure; Inflammation; Catecholamines
MeSH Terms: conditions — Inflammation | interventions — Psychological Tests; Vehicle Emissions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Filtered Air (No Intervention): Subjects sit in a room for two hours breathing in filtered air which resembles levels of air pollution found in the ambient environment
- Diesel Exhaust (Active Comparator): Subjects sit in a room for two hours breathing in diesel exhaust at 200 micrograms of meter cubed.
  Interventions: Other: Diesel exhaust
- TSST/Stress only (Active Comparator): Subjects undergo a mental stress test, known as the Trier Social Stress Test (TSST), which involves a public speaking and math task.
  Interventions: Behavioral: Trier social stress test
- Diesel Exhaust and stress (Active Comparator): Subjects sit in a room for two hours breathing in diesel exhaust at 200 micrograms of meter cubed and are subject to a mental stress test (TSST) which involves a public speaking and math task.
  Interventions: Behavioral: Trier social stress test; Other: Diesel exhaust

INTERVENTIONS:
Behavioral: Trier social stress test — Subjects are asked to give a 5 minute speech on a topic selected by the investigator. Then they are asked to subtract 7 from 758.
  Other Names: TSST
  Arms: Diesel Exhaust and stress; TSST/Stress only
Other: Diesel exhaust — Diesel exhaust is an air pollutant found in the environment and produced by cars, trucks and other transportation modes (e.g. trains, planes).
  Arms: Diesel Exhaust; Diesel Exhaust and stress

SUMMARY:
This study uses an experimental design to conduct a double-blind, randomized, crossover study where participants receive both diesel exhaust and a mental stress test in a controlled setting. My hypothesis is that the synergistic effect of stress and air pollution will result in higher levels of stress and inflammation (measured via biological markers) as well as poorer cardiovascular disease related outcomes compared to the independent effect of each exposure separately.

ELIGIBILITY:
Inclusion Criteria:

Non-smokers without history of high blood pressure, asthma, diabetes, high cholesterol, post-traumatic stress disorder (PTSD) or any other chronic condition that requires ongoing care.

Exclusion Criteria:

1. Smoking: We rule out active smoking by checking urine cotinine during our study.
2. History of high blood pressure: We objectively measure BP during in-person screening and exclude those with blood pressure (>130/85 mmHg).
3. Asthmatic: Spirometry is done at screening to rule out asthma.
4. Diabetic: We obtain fasting blood sugar to rule out diabetes at screening (>125 mg/dL)
5. Cholesterol: We obtain fasting blood lipid levels to rule out hypercholesterolemia at screening (>200 mg/dL).
6. History of PTSD: Subjects will be asked about prior PTSD diagnosis during the phone and in person screen.
7. Any other chronic condition requiring ongoing care based on medication use.
8. A body mass index (weight in kilograms divided by height in meters squared) greater than 26 and less than 18.5
9. A female of childbearing age with a positive pregnancy test
10. A female of childbearing age who is unwilling to use effective contraception during the study

Ages: 22 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Change in norepinephrine | Change in norepinephrine from baseline (pre-exposure) to immediately after exposure
  Urinary norepinephrine in ng/mg
Change in epinephrine | Change in epinephrine from baseline (pre-exposure) to immediately after exposure
  Urinary epinephrine in ng/mg
Change in dopamine | Change in dopamine from baseline (pre-exposure) to immediately after exposure
  Urinary dopamine in ng/mg

SECONDARY OUTCOMES:
Change in d-dimer | change in d-dimer from baseline (pre-exposure) to six hours post exposure
  plasma d-dimer (ug/ml) is a measure of coagulation
Change in fibrinogen | change in fibrinogen from baseline (pre-exposure) to six hours post exposure
  plasma fibrinogen (mg/dl) is a measure of coagulation
Change in interleukin-6 (IL-6) | change in IL-6 from baseline (pre-exposure) to immediately after exposure
  plasma IL-6, measured in pg/ml, is a marker of inflammation
Change in tumor necrosis factor alpha (TNF-a) | change in TNF-a from baseline (pre-exposure) to immediately after exposure
  plasma TNF-a, measured in pg/ml, is a marker of inflammation
Change in interleukin-1b (IL-1b) | change in IL-1b from baseline (pre-exposure) to immediately after exposure
  plasma IL-1b, measured in pg/ml, is a marker of inflammation

OTHER OUTCOMES:
Change in blood pressure | Change in blood pressure from baseline (pre-exposure) to 22 hours post exposure
  blood pressure in mm Hg
Change in heart rate | Change in blood pressure from baseline (pre-exposure) to 60 minutes post exposure
  heart rate in beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Anjum Hajat, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Diesel Exhaust Facility, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
We may share some of the clinical data collected such as blood pressure, spirometry and other markers of cardiac function with researchers interested in addressing related study questions. Direct identifiers will not be stored or shared, but rather only de-identified bio-specimens and data.